CLINICAL TRIAL: NCT05053347
Title: The Effect of Alpha Linolenic Acid Intake on Patients With Elevated Glycemic Status: a Double-blind Randomized Controlled Cross-over Trial
Brief Title: The Effect of Alpha Linolenic Acid Intake on Patients With Elevated Glycemic Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JWY20210916
Record Dates: First submitted 2021-09-16; First posted 2021-09-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Elevated Blood Sugar
MeSH Terms: conditions — Hyperglycemia | interventions — Linseed Oil; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flaxseed oil (Experimental): Flaxseed oil capsule, 4.5 g/d (ALA 2.5 g/d)
  Interventions: Dietary Supplement: Flaxseed oil capsule
- Corn oil (Placebo Comparator): Corn oil capsule, 4.5 g/d
  Interventions: Dietary Supplement: Corn oil capsule

INTERVENTIONS:
Dietary Supplement: Flaxseed oil capsule — The participants were asked to take flaxseed oil capsule 4.5 g/d (ALA 2.5g/d). The intervention period is 24 weeks separated by a 12-week washout period. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Flaxseed oil
Dietary Supplement: Corn oil capsule — The participants were asked to take corn oil capsule 4.5 g/d. The intervention period is 24 weeks separated by a 12-week washout period. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Corn oil

SUMMARY:
The findings of previous experiments suggested that alpha linolenic acid (ALA) has been linked to anti-hyperglycemic, and reducing the risk of diabetes.This is a randomized double-blind cross-over trial, aims to study the effect of ALA on glycemic status and human metabolism. Firstly, the investigators will investigate the efficacy of ALA on improving the indexes of glucose metabolism. Secondly, next generation sequencing (NGS), ultra-high performance liquid chromatography-tandem mass spectrometric (UPLC-MS/MS) and gas chromatography-mass spectrometry detection will be conducted to explore the role of ALA on gut microbiota as well as metabolites. Thirdly, single nucleotide polymorphism will be genotyped by Time-of-flight mass spectrometry to find the gene-environment interaction effect.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose 6.1-8.4mmol /L;
* HbA1c 5.7-7.0%;
* Patients with previously diagnosed type 2 diabetes with stable drug hypoglycemic treatment and blood glucose controlled well.

Exclusion Criteria:

* Under 30 years old or over 75 years old;
* Suffering from severe metabolic disorders, malignancies, psychiatric conditions;
* undergoing insulin therapy, or antibiotic/probiotic use for more than three consecutive days in the last month.
* Daily cooking oil is flaxseed oil, rapeseed oil or other α -linolenic acid rich vegetable oil;
* Intake more than 20g walnuts per day or more than 100g fatty fish per week in the last month;
* Take nutritional supplements, such as fish oil capsules, perilla seed oil and flaxseed oil capsules, for nearly one month;
* Allergic to the content of intervention;
* Failure to eat the tested sample as prescribed and affect the efficacy or safety judgment.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
changes of fasting blood glucose | 0 week, 12th week, 24th week and 36th week in the intervention period
  fasting blood glucose
changes of glycated hemoglobin (HbA1c) | 0 week, 12th week, 24th week and 36th week in the intervention period
  glycated hemoglobin (HbA1c)

SECONDARY OUTCOMES:
changes of circulating fatty acids | 0 week, 12th week, 24th week and 36th week in the intervention period
  plasma and erythrocyte fatty acid profiles
changes in the relative abundance of gut microbiota | 0 week, 12th week, 24th week and 36th week in the intervention period
  Evaluate alterations in the relative abundance of gut microbiota across taxonomic levels by 16S rRNA sequencing.
changes of fecal short-chain fatty acid | 0 week, 12th week, 24th week and 36th week in the intervention period
  fecal short-chain fatty acid
nutrient-gene interaction on circulating n-3 PUFAs | 0 week, 12th week, 24th week and 36th week in the intervention period
  The impact of genetic diversity in FADS and ELOVL gene clusters on changes in circulating n-3 PUFAs after ALA intervention.
nutrient-gene interaction on fasting blood glucose | 0 week, 12th week, 24th week and 36th week in the intervention period
  The impact of genetic diversity of diabetes-associated genes on changes in fasting blood glucose after ALA intervention.
nutrient-gene interaction on HbA1c | 0 week, 12th week, 24th week and 36th week in the intervention period
  The impact of genetic diversity of diabetes-associated genes on changes in HbA1c after ALA intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinopharm Dongfeng General Hospital, Shiyan, Hubei, China

IPD SHARING:
Plan to Share IPD: No